CLINICAL TRIAL: NCT06379854
Title: Effects Of Trunk Rotation And Lateral Flexion Exercises On Peak Cough Flow And Chest Expansion In Stroke Patients
Brief Title: Trunk Rotation And Lateral Flexion Exercises In Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCRAHS-ISB/REC/MS-PT/01814
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Stroke, Acute
Keywords: stroke; TRROM trunk rotation range of motion; TLFROM trunk lateral rotation range of motion; CPF cough peak flow meter
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chest physiotherapy (Experimental): we take 2 groups in one group only chest physiotherapy introduce
  Interventions: Other: chest physiotherapy
- trunk rotation exercises,deep diaphragmatic also chest physiotherapy (Active Comparator): But in 2nd group chest physiotherapy with trunk rotation exercises and deep diaphragmatic breathing exercises alo introduce.
  Interventions: Other: trunk rotation exercises,deep diaphragmatic also chest physiotherapy

INTERVENTIONS:
Other: chest physiotherapy — Postural Drainage Frequency: 3 sessions/week Intensity: 5 to 10 minutes Time: For 4 weeks Type: chest physiotherapy Percussion F: 3 sessions/week I: 3 to 5 minutes T: For 4 weeks T: chest physiotherapy Vibration F: 3 sessions/week I: 3 to 5 minutes T: For 4 weeks T: chest physiotherapy Shaking F: 3 sessions/week I: 3 to 5 minutes T: For 4 weeks T: chest physiotherapy Huffing and coughing F: 3 sessions/week I: 3 to 5 minutes T: For 4 weeks T: chest physiotherapy
  Arms: chest physiotherapy
Other: trunk rotation exercises,deep diaphragmatic also chest physiotherapy — Postural Drainage Frequency: 3 sessions/week Intensity: 5 to 10 minutes Time: For 4 weeks Type: chest physiotherapy
  Percussion F: 3 sessions/week I: 3 to 5 minutes T: For 4 weeks T: chest physiotherapy
  Vibration F: 3 sessions/week I: 3 to 5 minutes T: For 4 weeks T: chest physiotherapy
  Shaking F: 3 sessions/week I: 3 to 5 minutes T: For 4 weeks T: chest physiotherapy
  Huffing and coughing F: 3 sessions/week I: 3 to 5 minutes T: For 4 weeks T: chest physiotherapy
  Deep Diaphragmatic Breathing Exercise F: 3 sessions/week I: 3 to 5 minutes T: For 4 weeks T: chest physiotherapy TLFROM F: 3 sessions/week I: 5 to 10 minutes T: For 4 weeks T: Mobilization Exercises TFROM F: 3 sessions/week I: 5 to 10 minutes T: For 4 weeks T: Mobilization Exercises
  Arms: trunk rotation exercises,deep diaphragmatic also chest physiotherapy

SUMMARY:
In this study we want to introduce the beneficiary combine effects of chest mobilization and chest physiotherapy exercises by using cough peak flow meter and chest expansion in stroke patients. by using theses combine exercises physiotherapist can develop target rehabilitation strategies for stroke survivors.

DETAILED DESCRIPTION:
Stroke is a neurological deficit and acute focal injury of the by a vascular cause, including cerebral infarction, intracerebral hemorrhage and subarachnoid hemorrhage and is a major cause of disability and death worldwide. 2nd most deadly cause of death and disability in patients. This disease have long lasting effect on human body and also cause complication of lung function like pneumonia and respiratory distress function syndrome for this purpose to reduce chest complication and neurological defect use of chest physiotherapy and chest mobilization exercises are introduce so that hospital stay of patients reduces and recovery at high speed according to previous studies there is very strong relationship between trunk muscles and respiratory muscle with pulmonary function and physiotherapist can develop target rehabilitation strategies for stroke survivors.however in previous studies age group of patients acute subacute or chronic and diaphragmatic breathing are not included for the improvement of effective cough.

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* Age > 50
* Right or left hemiplegic acute stroke patients
* Diagnosed cases of stroke patient
* Duration: 4 weeks being diagnosed
* Can sit with at least 10sec
* Can perform exercises with Active Assistance
* Patients who easily perform exercises
* Patients who response to commands

Exclusion Criteria:

* Patients with serious comorbidities like cancer
* Uncontrolled hypertension SBP > 140mmhg and DBP > 90mmhg
* Vitally unstable patient's
* Red flags for physiotherapy i.e. sudden dizziness, unexplained pain during exercise, chest pain.
* DVT Deep Vein Thrombosis

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Trunk Impairment Scale: | 4th week
  Changes from baseline this scale is used to assess motor impairment of the trunk after stroke through the evaluation of static and dynamic sitting balance as well as coordination of trunk movement. The initial static sitting balance score 0 means overall total score is O. and full score is 23. This tool is also used to assess progress of trunk movement.
Peak Flow Meter | 4th week
  Changes from baseline Peak flow meter is used to access the peak cough flow in stroke patient's pre and post intervention. Cough peak flow (CPF) measures the maximum expiratory flow during the phase of a cough just after instant opening of the glottis, but peak expiratory flow rate (PEFR) measures maximum expiratory flow, after a full deep inspiration, through an open glottis Normal peak cough flow is about greater than or equal to 270L/min. And the ineffective cough is about less than 160L/min.
Chest Expansion: | 4th week
  A tape measure is used to evaluate the both upper and lower chest expansion in stroke patients. These chest expansions were performed three time and mean value of these are taken. By using tape measure, we determine the difference between rib cage circumference at the end of forced inspiration and at the end of forced expiration. The reliability score for chest expansion is about (0.99)

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, phd*, Principal Investigator — Riphah International University
Locations (1):
- Shahida Khaliq Health Centre, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sacco RL, Kasner SE, Broderick JP, Caplan LR, Connors JJ, Culebras A, Elkind MS, George MG, Hamdan AD, Higashida RT, Hoh BL, Janis LS, Kase CS, Kleindorfer DO, Lee JM, Moseley ME, Peterson ED, Turan TN, Valderrama AL, Vinters HV; American Heart Association Stroke Council, Council on Cardiovascular Surgery and Anesthesia; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular and Stroke Nursing; Council on Epidemiology and Prevention; Council on Peripheral Vascular Disease; Council on Nutrition, Physical Activity and Metabolism. An updated definition of stroke for the 21st century: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2013 Jul;44(7):2064-89. doi: 10.1161/STR.0b013e318296aeca. Epub 2013 May 7. PMID 23652265
- [Background] Johnson W, Onuma O, Owolabi M, Sachdev S. Stroke: a global response is needed. Bull World Health Organ. 2016 Sep 1;94(9):634-634A. doi: 10.2471/BLT.16.181636. No abstract available. PMID 27708464
- [Background] Saini V, Guada L, Yavagal DR. Global Epidemiology of Stroke and Access to Acute Ischemic Stroke Interventions. Neurology. 2021 Nov 16;97(20 Suppl 2):S6-S16. doi: 10.1212/WNL.0000000000012781. PMID 34785599
- [Background] Turana Y, Tengkawan J, Chia YC, Nathaniel M, Wang JG, Sukonthasarn A, Chen CH, Minh HV, Buranakitjaroen P, Shin J, Siddique S, Nailes JM, Park S, Teo BW, Sison J, Ann Soenarta A, Hoshide S, Tay JC, Prasad Sogunuru G, Zhang Y, Verma N, Wang TD, Kario K; HOPE Asia Network. Hypertension and stroke in Asia: A comprehensive review from HOPE Asia. J Clin Hypertens (Greenwich). 2021 Mar;23(3):513-521. doi: 10.1111/jch.14099. Epub 2020 Nov 15. PMID 33190399
- [Background] Farooq A, Venketasubramanian N, Wasay M. Stroke Care in Pakistan. Cerebrovasc Dis Extra. 2021;11(3):118-121. doi: 10.1159/000519554. Epub 2021 Oct 25. PMID 34695824
- [Background] Yew KS, Cheng EM. Diagnosis of acute stroke. Am Fam Physician. 2015 Apr 15;91(8):528-36. PMID 25884860
- [Background] Rochester CL, Mohsenin V. Respiratory complications of stroke. Semin Respir Crit Care Med. 2002 Jun;23(3):248-60. doi: 10.1055/s-2002-33033. PMID 16088617
- [Background] Jeong, J.-H., Brain and lung: lung injury in patients with brain injury. Journal of Neurocritical Care, 2017. 10(1): p. 1-6.
- [Background] Kim, A., et al., Effects of rib cage joint mobilization combined with diaphragmatic breathing exercise on the pulmonary function and chest circumference in patients with stroke. Journal of International Academy of Physical Therapy Research, 2020. 11(3): p. 2113-2118.
- [Background] Belal, E.S., S. Selim, and A. Mohammad, Detection of airway protective level of the cough reflex in acute stroke patients. The Egyptian Journal of Neurology, Psychiatry and Neurosurgery, 2020. 56(1): p. 1-6.
- [Background] Park, S.J., Effects of inspiratory muscles training plus rib cage mobilization on chest expansion, inspiratory accessory muscles activity and pulmonary function in stroke patients. Applied Sciences, 2020. 10(15): p. 5178.
- [Background] Khedr EM, El Shinawy O, Khedr T, Aziz Ali YA, Awad EM. Assessment of corticodiaphragmatic pathway and pulmonary function in acute ischemic stroke patients. Eur J Neurol. 2000 May;7(3):323-30. doi: 10.1046/j.1468-1331.2000.00078.x. PMID 10886317
- [Background] Verheyden G, Nieuwboer A, De Wit L, Feys H, Schuback B, Baert I, Jenni W, Schupp W, Thijs V, De Weerdt W. Trunk performance after stroke: an eye catching predictor of functional outcome. J Neurol Neurosurg Psychiatry. 2007 Jul;78(7):694-8. doi: 10.1136/jnnp.2006.101642. Epub 2006 Dec 18. PMID 17178824
- [Background] Waseem, M.H., et al., Effectiveness of chest physiotherapy in cerebrovascular accident patients with aspiration pneumonia. Journal of Modern Rehabilitation, 2021. 15(1): p. 47-52.
- [Background] Jang SH, Bang HS. Effect of thoracic and cervical joint mobilization on pulmonary function in stroke patients. J Phys Ther Sci. 2016 Jan;28(1):257-60. doi: 10.1589/jpts.28.257. Epub 2016 Jan 30. PMID 26957769
- [Background] Park HY, Hwang UJ, Kwon OY. Correlation between trunk rotation and lateral flexion range of motion, peak cough flow, and chest expansion in stroke patients. Physiother Res Int. 2023 Jan;28(1):e1970. doi: 10.1002/pri.1970. Epub 2022 Aug 12. PMID 35962597
- [Background] Messaggi-Sartor M, Guillen-Sola A, Depolo M, Duarte E, Rodriguez DA, Barrera MC, Barreiro E, Escalada F, Orozco-Levi M, Marco E. Inspiratory and expiratory muscle training in subacute stroke: A randomized clinical trial. Neurology. 2015 Aug 18;85(7):564-72. doi: 10.1212/WNL.0000000000001827. Epub 2015 Jul 15. PMID 26180145
- [Background] Jo, M.-R., N.-S. Kim, and J.-H. Jung, The effects of respiratory muscle training on respiratory function, respiratory muscle strength, and cough capacity in stroke patients. Journal of Korean Society of Physical Medicine, 2014. 9(4): p. 399-405.